CLINICAL TRIAL: NCT05720403
Title: The Effect of Pilates in Pregnant Women: A Randomized Controlled Study
Brief Title: Investigation of the Effects of Pilates Training in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Bulguroglu, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Healthy Lifestyle; Health Behavior
Keywords: Pilates exercises; Pregnant; Mood; Core
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Using a computer program, the investigators randomly placed individuals who completed the initial assessment into the pilates group (PG) or control group (CG).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were evaluated at the beginning of the study and 8 weeks later by an experienced physical therapist blind to randomization. The group participants belonged to was not disclosed to the participants from the initial assessment to the end.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates group (Experimental): Pilates, which lasts for eight weeks, three days a week for 1 hour, will be carried out by Australian Pilates and Physiotherapy Institute certified and experienced Ph.D. Physiotherapist Halil Ibrahim Bulguroglu. The individuals in pilates exercise groups will be divided into six small groups to make the exercises more effective. In this study, the program will be 15 minutes of warm-up, 30 minutes of pilates, and 15 minutes cool-down and stretching exercises. The exercises will be performed in ten repetitions.
  Interventions: Other: pilates group
- control group (No Intervention): The group received breathing and relaxation exercises with a home program.

INTERVENTIONS:
Other: pilates group — Pilates, which lasts for eight weeks, three days a week for 1 hour, will be carried out by Australian Pilates and Physiotherapy Institute certified and experienced Ph.D. Physiotherapist Halil Ibrahim Bulguroglu. Microsoft Teams program will be used to implement the online practice method. The individuals in both pilates exercise groups will be divided into six small groups of 3 or 4 people to make the exercises more effective. In this study, the program will be 15 minutes of warm-up, 30 minutes of pilates, and 15 minutes of cool-down and stretching exercises. The exercises will be performed in ten repetitions. The same exercises will be applied in online pilates and face-to-face pilates training.
  Arms: pilates group

SUMMARY:
Pregnancy is a physiological stress state that affects all body systems and requires physical, mental, and social harmony in the woman.

The pregnancy process continues with visible changes in the female body and psychological changes and fluctuations. The mental and physical adaptation of the mother to the changes that occur during pregnancy can be increased by interventions that can be done in this process. Exercises are at the top of these interventions.

Exercise has been shown to affect the fetus, mother, and pregnancy positively. In the guide published by the American Obstetricians and Gynecologists Committee in 2015, It was stated that pregnant women should exercise at least half an hour of moderate-intensity on most days of the week. They also recommended exercises such as Pilates, yoga, and swimming as safe activities for pregnant women.

Pilates exercises are ideal for preparing the pregnant woman's body until birth, and after birth plays a vital role in the recovery of the mother's body. Above all, it makes women feel more comfortable in this temporary body and makes them more active. When the literature is examined, it is seen that studies which include the effects of Pilates during pregnancy are still insufficient All of these studies examining the effects of Pilates education on pregnant women show us that Pilates education can positively contribute to pregnant women. However, in all studies, it is stated that the effects of Pilates on different dimensions of pregnancy should be examined, and additional studies with high evidence value are needed.

Based on this, to ensure that pregnant women have a healthier and more comfortable pregnancy period, a randomized controlled blind study was planned to investigate the effects of Pilates training on core stability, balance, mood, and quality of life in pregnant women.

DETAILED DESCRIPTION:
Pilates exercises are ideal for preparing the pregnant woman's body until birth and after the delivery and play a vital role in the recovery of the mother's body. Above all, it makes women feel more comfortable in this temporary body and causes them to be more active. When the literature is examined, it is seen that studies which include the effects of Pilates during pregnancy are still insufficient. All of these studies examining the impact of Pilates education on pregnant women show us that Pilates education can positively contribute to pregnant women. However, in all studies, it is stated that the effects of Pilates on different dimensions of pregnancy should be examined, and additional studies with high evidence value are needed.

Based on this, to ensure that pregnant women have a healthier and more comfortable pregnancy period, a randomized controlled blind study was planned to investigate the effects of Pilates training on core stability, balance, mood, and quality of life in pregnant women.

Fifty-eight pregnant women, who completed the first trimester of pregnancy, have been included in the study. Inclusion and exclusion criteria were established according to the guidelines of the American Obstetricians and Gynecologists Committee. The Local Ethics Committee approved the study and written informed consent was obtained from all patients to participate.

- Procedures The subjects were separated into two groups, Pilates and the control group, in a randomized manner. The Pilates method was given by a physiotherapist with an Australian Pilates and Physiotherapy Institute certificate and was experienced in pregnancy and Pilates. The control group was followed through the home program. The blind physiotherapist did the evaluations before and after the treatment.

Pilates groups were taken into about one hour of training two days a week. Pregnancy training exercises recommended by the Australian Pilates and Physiotherapy Institute were used in training. Throughout the Pilates training, the physiotherapist controlled the movements, and the necessary corrections were made through tactile and verbal warnings and imagery. The subjects in the control group were asked to follow a home program that consisted of relaxation and respiration exercises for eight weeks, two times per week.

Core stability, balance, mood, and quality of life were evaluated before and after the study.

In our study, it was thought that the application of all core stability tests in pregnant women may not be appropriate for the safety of pregnant women and that pregnancy is a factor affecting the reliability of the test. Therefore, the Sahrmann core stability test and core endurance tests evaluated core stability. Among the core endurance tests, trunk flexion test, right-left side bridge test, and prone bridge test were used.

Sharman Core Stability Test: Consists of 5 levels. Level 1 was applied to pregnant women. The pregnant woman was laid on her back and knees flexed for the test. The biofeedback device (Stabilizer™, Chattanooga Group Inc., Chattanooga, TN) was placed in the lumbar region. Then the pressure biofeedback was inflated to 40 mmHg. In this position, the abdominal draw-in maneuver was taught, which provides remote activation of M. transversus abdominis. The pregnant were asked to flex their legs one by one and then both. The pressure change in the device during the test was recorded.

Core endurance measurements were recorded with a clock as seconds. The tests ended when the subjects broke the test positions.

Side bridge test: The subjects were asked to lay on their left or right sides and to extend their legs entirely. Then the subjects were asked to create a straight line with their body by lifting their hip from the floor.

Trunk flexion test: This was initiated when the subjects sat up with their back resting against a wedge angled 55◦ from the floor.

Prone bridge test: In this test, the subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight as they are required not to arch or bow.

Balance was evaluated using the Biodex-BioSway™ (Biodex Medical Systems, Shirley, NY, USA) Portable Balance System, an objective measurement method. This device assesses balance with three different tests. In our study, a postural stability test was used. This test evaluates the individual's ability to hold the center of gravity on the support surface during standing. In our study, total stability index scores of the right, left, and double legs were used for statistical analysis.

Three different questionnaires evaluated the moods of the pregnant. Edinburgh Postnatal Depression Scale (EPDS): In 2009, it was stated that EPDS was a reliable tool for assessing depressive symptoms during pregnancy. The scale is a self-report scale consisting of 10 items.

The Wijma Delivery Expectancy/Experience Scale- A version (W-DEQ A) was developed to measure the fear of birth. The 33-item scale is a six-point Likert-type scale.

State-Trait Anxiety Scale (STAI Form 1-2): The Likert-type scale measures state and trait anxiety levels separately with 20 questions.

Quality of life was evaluated with Short Form-36. The scale consists of 36 items and provides the measurement of 8 dimensions. The fourth and fifth questions of the scale are considered with yes/no, and the other questions are reviewed with a Likert-type rating.

Statistical Analysis SPSS 21.0 (SPSS Inc., Chicago, IL, USA) for Windows software program was used in all statistical analyses. In the data evaluation, mean, standard deviation, median, interquartile range, and minimum and maximum values were used for numerical measurements among descriptive statistics. Whether measurements display normal distribution was tested with the Shapiro-Wilk test. The Mann-Whitney u test and Independent Samples T-test were performed in the two-group comparisons. A p<0.05 was accepted as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years of age
* Voluntarily participate in research to accept
* 12-28 weeks of pregnancy
* Singleton pregnancy

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing, and perception problems may affect the research results.
* Participating in other exercises or physiotherapy programs during the past six months.
* Multiple pregnancies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Core Stability Test- Baseline | Assessment will be conducted before the intervention
  Sahrman Core Stability Test
Core Stability Test-Post intervention | Assessment will be conducted immediately after the intervention
  Sahrman Core Stability Test
Balance - Baseline | Assessment will be conducted before the intervention
  Balance was evaluated using the Biodex-BioSway™ (Biodex Medical Systems, Shirley, NY, USA) Portable Balance System
Balance - Post intervention | Assessment will be conducted immediately after the intervention
  Balance was evaluated using the Biodex-BioSway™ (Biodex Medical Systems, Shirley, NY, USA) Portable Balance System
Quality of life - Baseline | Assessment will be conducted before the intervention
  Short Form-36 (SF-36). SF-36; consists of 36 items to measure eight dimensions such as physical, mental, and general health. In the subscales evaluated between 0 and 100, a high score indicates a good quality of life.
Quality of life - Post intervention | Assessment will be conducted immediately after the intervention
  Short Form-36 (SF-36). SF-36; consists of 36 items to measure eight dimensions such as physical, mental, and general health. In the subscales evaluated between 0 and 100, a high score indicates a good quality of life.
Fear of Birth- Baseline | Assessment will be conducted before the intervention
  The Wijma Birth Expectation/Experience Scale was developed to measure the nature of the fear of childbirth during and after labor by asking women questions about their experiences after birth. The minimum score on the scale is 33, and the maximum score is 198
Fear of Birth- Post intervention | Assessment will be conducted immediately after the intervention
  The Wijma Birth Expectation/Experience Scale was developed to measure the nature of the fear of childbirth during and after labor by asking women questions about their experiences after birth. The minimum score on the scale is 33, and the maximum score is 198

CONTACTS AND LOCATIONS:
Overall Officials: HALİL İ BULGUROGLU, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Altındağ, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Mazzarino M, Kerr D, Morris ME. Pilates program design and health benefits for pregnant women: A practitioners' survey. J Bodyw Mov Ther. 2018 Apr;22(2):411-417. doi: 10.1016/j.jbmt.2017.05.015. Epub 2017 May 31. PMID 29861243
- [Result] Satyapriya M, Nagendra HR, Nagarathna R, Padmalatha V. Effect of integrated yoga on stress and heart rate variability in pregnant women. Int J Gynaecol Obstet. 2009 Mar;104(3):218-22. doi: 10.1016/j.ijgo.2008.11.013. Epub 2008 Dec 25. PMID 19110245
- [Result] Barakat R, Cordero Y, Coteron J, Luaces M, Montejo R. Exercise during pregnancy improves maternal glucose screen at 24-28 weeks: a randomised controlled trial. Br J Sports Med. 2012 Jul;46(9):656-61. doi: 10.1136/bjsports-2011-090009. Epub 2011 Sep 26. PMID 21948120